CLINICAL TRIAL: NCT04117594
Title: Whole Body Magnetic Resonance Imaging Study
Acronym: WISE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5035
Record Dates: First submitted 2019-09-26; First posted 2019-10-07 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Advanced Prostate Cancer
Keywords: Prostate cancer; WB-MRI; Bone disease
MeSH Terms: conditions — Prostatic Neoplasms; Bone Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: WB-MRI — Whole body MRI with diffusion-weighted imaging (DWI)

SUMMARY:
In prostate cancer bone is the most common site for cancer spread, causing pain, fractures, nerve compression and death.

New therapies are available for treating bone disease from cancer and this means that by maintaining patients on drugs that are effective and switching patients to other drugs when current treatment becomes ineffective, patients can be maintained 'better for longer'. However, to do this, it is necessary to accurately tell whether a given treatment is working or not.

In this study, the investigators will perform whole body MRI scans, which include a special scan called diffusion-weighted MRI (DWI MRI) that can provide more information about the participants extent of disease. The investigators aim to show that this test is better than the standard tests of CT and bone scan currently used in the NHS to monitor bone disease. The information from this study will be used to test a special software so that the test may more widely benefit patients across the NHS in the future.

DETAILED DESCRIPTION:
In patients with prostate cancer the current methods to assess treatment response of bone disease such as computer tomography (CT) and bone scan (BS)are unreliable, insensitive to bone disease and have limited criteria to assess disease response confined to bones. Blood tests are inaccurate although some newer tests (e.g. circulating tumour cells tests) show promise but are still under investigation and nuclear medicine investigations such as PET/CT imaging have higher sensitivity, meaning they can detect more sites of disease who are indeed disease than CT or BS but they are more costly and less widely available compared with MRI within the NHS.

For this study the Whole body MRI (WB-MRI) includes a measurement called diffusion-weighted imaging (DWI) which is relatively new and has a high sensitivity for bone metastases. This technique can be used to measure total bone disease volume (TDV) and the disease apparent diffusion coefficient (ADC) which reflects the tumour tissue cell density. Previous studies have shown good reproducibility of both these measurements and a significant increase in the mean tumour ADC is observed in patients who are responding to effective treatment.

However WB-MRI application across the NHS is ad-hoc, CT and BS techniques are entrenched within clinical practice despite their known limitations. Another factor that limits wider adoption of WB-MRI is the lack of sophisticated analysis software to enable disease across the body to be quickly evaluated.

This multi-centre imaging study will provide the opportunity to evaluate the performance of WB-MRI with a novel software diagnostics for evaluating the treatment response of advanced prostate cancer patients.

This prototype can used to evaluate WB-MRI data from different scanners and address a current major unmet need for the treatment and follow-up of patients with bone disease from cancers, so that the test may more widely benefit patients across the NHS in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥18 years
3. Patients with APC with predominantly bone disease confirmed by bone scan (within 6 weeks) or CT (within 6 weeks), of starting treatment (Cycle 1 Day 1). Patients with local recurrence and bone metastases with an associated soft tissue component, will be allowed into the trial. Pelvic lymphadenopathy <1.5cm in short axis is not an exclusion.
4. Systemic therapy indicated for disease progression, as clinically indicated.

Exclusion Criteria:

1. Patient is claustrophobic.
2. Contraindications to MRI examination (e.g. cardiac pacemakers, cochlear implants).
3. Measurable soft tissue or lymph node metastases or any metastatic disease outside the bone that is RECIST measurable will be an exclusion (unless it is pelvic nodal disease <1.5cm in short axis). Bone metastases with associated soft tissue components will also not be an exclusion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with advanced prostate cancer
Study Population: Advanced prostate cancer patients with bone predominant metastases and no RECIST-measurable disease (lymph nodes <1.5cm in short axis in the pelvis are allowed) who have an indication for systemic treatment (taxane chemotherapy or AR targeted agents).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of WB MRI at post treatment by quantification of bone disease | End of Cycle 3 of treatment (each cycle being 28 days or 21 days depending on the type of standard therapy)
  To establish the diagnostic performance of whole body MRI (WB MRI) using total bone disease volume (TDV) and disease apparent diffusion coefficient (ADC) at Cycle 3 (within 2 weeks before treatment on C4 Day1, each cycle being 28 days or 21 days depending on the type of standard therapy) using new software diagnostics for assessing treatment response to standard therapy (taxane chemotherapy or AR targeted agents)) in patients with bone predominant metastatic disease in prostate cancer using a construct reference standard.

SECONDARY OUTCOMES:
Compare diagnostic performance of WB-MRI at Cycle 3 versus standard imaging CT and bone scan by quantification of bone disease | End of Cycle 3 of treatment (each cycle being 28 days or 21 days depending on the type of standard therapy)
  Compare the diagnostic performance of WB-MRI using TDV and ADC at Cycle 3 (within 2 weeks before treatment on C4 Day1, each cycle being 28 or 21 days depending on the type of standard therapy) with the diagnostic performance of standard imaging CT and BS (when available).
Time to progression of responders and non-responders | 6 months
  Determine the time to progression of responders and non-responders to therapy as defined by WB MRI, versus CT and BS.
Intra-observer and inter-observer agreement of ADC and TDV | 1 year
  Assess the intra-observer and inter-observer agreement of the apparent diffusion coefficient (ADC) and total diffusion volume (TDV) of bone disease assessed by WB-MRI.
Assess the cost-effectiveness of replacing CT and BS with WB-MRI derived measurements TDV and ADC | 1 year
  Determine the cost-effectiveness of replacing CT and BS with WB-MRI derived TDV and ADC measurements for disease management in patients with prostate bone disease using QALYs.

OTHER OUTCOMES:
Histogram parameters of ADC | 6 months
  Explore histogram parameters of ADC in responders and non-responders to treatment.
Histogram parameters of TDV | 6 months
  Explore histogram parameters of TDV in responders and non-responders to treatment.
Histogram parameters of fat fractions | 6 months
  Explore histogram parameters of fat fractions in responders and non-responders to treatment.
Cost and cost-effectiveness to the NHS of replacing the standard practice conventional tests | 1 year
  Assess the cost and cost-effectiveness to the NHS of replacing the standard practice conventional tests CT and BS with WB-MRI-derived TDV and ADC measurements for disease management in patients with prostate bone disease using the advanced computer diagnostics software in development using QALYs and obtained from survival data and health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised trial data will be made available
Supporting Information: CSR
Time Frame: Data will be available within 1 year of study completion.